CLINICAL TRIAL: NCT05770882
Title: A Phase Ib/II, Two-part, Non-randomized, Open-label Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Chidamide in Combination With Regorafenib in Patients With Hepatocellular Carcinoma
Brief Title: Chidamide + Regorafenib in Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The overall profile does not support development for Hepatocellular Carcinoma
Sponsor: Great Novel Therapeutics Biotech & Medicals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KEPIDA-1
Record Dates: First submitted 2023-02-07; First posted 2023-03-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; HBI-8000; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Part I safety; and Part II cohort expansion (Experimental): Part I: The safety of drug combination will be studied.
  Part II: The drug combination will be further evaluated in the cohort expansion phase.
  Interventions: Drug: Chidamide; Drug: Regorafenib

INTERVENTIONS:
Drug: Chidamide — Subjects will receive a single dose of chidamide. 5mg tablet. One dose every three days.
  Other Names: Tucidinostat; HBI-8000
Drug: Regorafenib — Subjects will receive a single dose of Regorafenib. 40mg tablet. One dose daily.
  Other Names: Stivarga; BAY 73-4506

SUMMARY:
This open-label, phase Ib/II, multicenter study evaluated the safety, tolerability, efficacy, and PK of chidamide in combination with regorafenib in patients with HCC. Chidamide, a histone deacetylase inhibitor, functions as a tumor inhibitor. Regorafenib, a receptor tyrosine kinase inhibitor, was approved as second-line systemic treatment for HCC patients.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase Ib/II study, which includes a Part I (phase Ib) and a Cohort Expansion part (Part II; phase II). Part I of the study is designed to assess the safety, tolerability, PK profiles, efficacy, and PD biomarkers of the study medications in patients with HCC. Part II of the study is designed to assess the efficacy, safety, and PD biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of HCC or non-invasive diagnosis of HCC as per American Association for the Study of Liver Diseases (AASLD) criteria in patients with a confirmed diagnosis of cirrhosis.
2. Barcelona Clinic Liver Cancer (BCLC) stage B or C HCC that cannot benefit from treatments of established efficacy with higher priority such as resection, local ablation, chemoembolization or first-line systemic therapy.
3. Has received and failed one front-line systemic treatment with either sorafenib, lenvatinib, or combination of PD-1/PD-L1 immune checkpoint inhibitor (ICI; anti-PD-1/PD-L1 mAb) plus bevacizumab, lenvatinib or anti-CTLA-4 mAb.
4. Tolerability of prior treatment with sorafenib or lenvatinib. Tolerability to previous sorafenib treatment is defined as not less than 20 days at a minimum daily dose of 400 mg QD within the last 28 days prior to withdrawal. Tolerability to previous lenvatinib treatment is defined as not less than 20 days at a daily dose of 8 mg QD for patients ≥60 kg or 4 mg QD for patients <60 kg days within the last 28 days prior to withdrawal.
5. Liver function status Child-Pugh Class A. Child-Pugh status should be calculated based on clinical findings and laboratory results during the screening period.
6. Local or loco-regional therapy of intrahepatic tumor lesions (e.g., surgery, radiation therapy, hepatic arterial embolization or infusion chemotherapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) must have been completed ≥4 weeks before the first dose of study medication.
7. ECOG PS of 0 or 1.
8. With adequate bone marrow, liver, and renal functions, as assessed by the following laboratory tests conducted within 7 days before the first dose of study medication:
9. At least one uni-dimensional measurable lesion by computed tomography scan or magnetic resonance imaging according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and modified RECIST for HCC (mRECIST). Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, may be considered measurable if there has been demonstrated progression in the lesion.
10. With a life expectancy of at least 3 months.
11. Females of childbearing potential and males must agree to use adequate contraception since signing of the informed consent form until at least 2 months after the last study drug administration.
12. Female patients of childbearing potential must have a negative urine or serum pregnancy test.
13. Able to take oral medication.
14. Has ability to understand and the willingness to provide a written informed consent document.

Exclusion Criteria:

1. With history of organ transplantation or candidates for liver transplantation.
2. Prior treatment with regorafenib.
3. First-line treatment within 4 weeks before the first dose of study medication.
4. Permanent discontinuation of prior sorafenib or lenvatinib therapy due to drug-related toxicity.
5. Known history or symptomatic metastatic brain or meningeal tumors. Note: If patients showed symptomatic brain metastases at screening, magnetic resonance imaging (MRI) or computed tomography (CT) scanning should be performed to demonstrate any current evidence of progressive brain metastases.
6. Major surgical procedure or significant traumatic injury within 28 days before the first dose of study medication.
7. With uncontrolled or significant cardiovascular diseases
8. With the size of fluid area detected by cardiac ultrasonography in cavum pericardium ≥ 10 mm.
9. Patients with pheochromocytoma.
10. Uncontrolled ascites (defined as not easily controlled with diuretic or paracentesis treatment).
11. Pleural effusion or ascites that causes respiratory compromise (National Cancer Institute - Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0 grade ≥2 dyspnea).
12. Ongoing infection grade >2 according to NCI-CTCAE v5.0. Hepatitis B is allowed if no active replication is present. Hepatitis C is allowed if no antiviral treatment is required.
13. Clinically significant bleeding NCI-CTCAE v5.0 grade ≥3 within 30 days before the first dose of study medication.
14. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months before the first dose of study medication..
15. With autoimmune disorders or history of organ transplantation who require immunosuppressive therapy
16. Non-healing wound, ulcer, or bone fracture.
17. Renal failure requiring hemo- or peritoneal dialysis.
18. Interstitial lung disease with ongoing signs and symptoms at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) | From the first day of treatment until progressive disease or death, assessed up to 12 months
  To analyze the frequency, percentage of patients with study medications of adverse events
Maximum tolerated dose(MTD) / maximum feasible dose (MFD) | From start of treatment Cycle1 Day1 until completion of one cycle of treatment (maximum 28 days)
  To assess tolerability/feasible of study medications dose
Pharmacokinetics profiles - (AUC0-t) | Blood samples collected on Days 1-4 and 18-21 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Area under the plasma concentration-time curve from time zero to time t(AUC0-t)
Pharmacokinetics profiles - (AUC0-∞) | Blood samples collected on Days 1-4 and 18-21 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Area under the plasma concentration-time curve from time zero to infinity(AUC0-∞)
Pharmacokinetics profiles - (Cmax) | Blood samples collected on Days 1-4 and 18-21 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Maximum plasma concentration(Cmax)
Pharmacokinetics profiles - (Tmax) | Blood samples collected on Days 1-4 and 18-21 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Time to maximum plasma concentration(Tmax)
Pharmacokinetics profiles - (T1/2) | Blood samples collected on Days 1-4 and 18-21 of Cycle 1, pre-dose and up to 72 hours post-dose (28 days/cycle)
  Half-life(T1/2)
Objective response rate (ORR) | Objective Response Rate is assessed every 8 weeks from start of treatment until progressive disease is documented (approximately 6 months)
  The percentage of patients with CR and PR of total number of analysis set
Progression-free survival (PFS) | From the first day of treatment until disease progression or death from any cause, assessed up to 12 months
  The time from first day of dosing until the date of first objective disease progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year
  The time from the first day of dosing until the date of death
Time to progression (TTP) | 1 year
  The time from the first day of dosing until the date of progression

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Nan Chen, Ph.D., Study Director — Great Novel Therapeutics Biotech & Medicals Corporation
Locations (5):
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided